CLINICAL TRIAL: NCT03273673
Title: Reduction of Risk Factors for ACL Re-injuries Using an Innovative Biofeedback Approach
Brief Title: Reduction of Risk Factors for ACL Re-injuries Using a Novel Biofeedback Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Robin Queen, Associate Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-007; R21AR069865-01A1 (NIH)
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Results first posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: Secondary ACL Injury Prevention; Visual Biofeedback; Tactile Biofeedback
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: This study involves one active intervention group and an attention control group
Who Masked: Care Provider, Outcomes Assessor
Masking Description: To reduce the possibility of bias, the biofeedback intervention will be completed by a single individual (clinician - Athletic trainer) and the biomechanical assessments will be completed by a second individual who will be blinded to the subject's group assignment (research technician).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback Intervention (Experimental): The 6-week biofeedback training program is focused on altering loading and movement asymmetry during biweekly sessions on non-consecutive days (12 sessions). The biofeedback training program will provide sensory (visual and tactile) feedback to the subject to heighten awareness of asymmetrical movement strategies (e.g. load shift, movement asymmetry) during a squat. The two exercises that will be completed during the biofeedback training program will be a visual feedback squat and a resisted squat (tactile feedback). Each of these tasks will be completed 30 (3 sets of 10 repetitions) times per session. We will provide a 20 second rest between trials, and a 10 minute break between the visual and tactile feedback exercises to decrease the effect of fatigue.
  Interventions: Other: Biofeedback Intervention
- Control (No Intervention): The 6-week attention control group program will focus on providing educational information to the participants related to the clinical and sports expectations as they are released to return to sport. These participants will be asked to meet 6 times during the 6-week intervention time period. Three of these visits will be completed in person and three will be completed using an online educational module (6 sessions). The online sessions will be completed in week 1, week 3, and week 5 while the in person sessions will be completed during week 2, week 4, and week 6.

INTERVENTIONS:
Other: Biofeedback Intervention — Visual and Tactile Biofeedback
  Arms: Biofeedback Intervention

SUMMARY:
ACL injuries are common among athletes and due to residual muscle weakness, limited knee motion and asymmetrical movement patterns after surgery many of these athletes will sustain secondary ACL injuries following return to sports. This project seeks to determine if a novel biofeedback-based rehabilitation approach can decrease a known risk factor for secondary injuries to the ACL. The project specifically focuses on correcting asymmetric movement patterns, a known risk factor for secondary injury that is not directly addressed by existing interventions through a 6 week therapy based biofeedback intervention.

DETAILED DESCRIPTION:
Nearly 1 in 60 adolescent athletes will suffer ACL injuries. Approximately 90% of these injured athletes will undergo an ACL reconstruction at an estimated annual cost of $3 billion. While reconstruction and subsequent rehabilitation allow these athletes to return to sports, they have a 15 fold increased risk of secondary ACL injuries, a tear of the ACL graft or the contralateral ACL. As a result, development of an intervention to reduce the incidence of secondary ACL tears would meet a critical need. One area in which existing interventions might be improved is through an increased emphasis on correcting asymmetric movement patterns-a known risk factor for secondary injury. Thus, our long-term objective is to decrease the number of secondary ACL tears by decreasing side-to-side movement and loading asymmetry. The modification of post-operative rehabilitation to focus on movement and loading symmetry with shift the rehabilitation paradigm. Specifically, we propose to evaluate a novel biofeedback training program that focuses on altering loading and movement patterns to improve symmetry and overall lower extremity mechanics in a group of 40 (20 control, 20 intervention) adolescent ACL reconstructed patients. There are two core hypotheses of this study: 1) biofeedback training will decrease known risk factors for secondary ACL injuries immediately following the biofeedback program and these changes will be retained 6 week after the completion of the biofeedback program; and 2) we will be able to recruit and enroll 40 patients and retain 80% of the patients through the end of the follow-up assessment demonstrating the feasibility of the biofeedback intervention. Implementation of a biofeedback program prior to returning to dynamic athletic activities could improve physical performance outcomes, decrease secondary injury risk factors and ultimately decrease the long-term joint degeneration and development of osteoarthritis that has been associated with ACL reconstruction. Ultimately this work will lead to additional investigations to definitively determine the impact of this novel biofeedback program, which could shift the post-operative rehabilitation paradigm following ACL reconstruction to improve long-term joint health in these adolescent patients.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. ACL Reconstruction: primary, unilateral ACL reconstruction with no pain in the contralateral leg
3. Rehabilitation: need to have completed at least 4.5 months of post-operative physical therapy and be within approximately 6 weeks of being ready to be released by his/her treating orthopaedic surgeon to return to full sport participation
4. Stated willingness to comply with all study procedures and availability for the duration of the study
5. Male or female, aged 14-21
6. Willing to adhere to the ACL Biofeedback intervention regimen

Exclusion Criteria:

1. For females: currently pregnant or planning to become pregnant
2. History of more than one ACL reconstruction
3. Post-operative complications that required additional surgical intervention
4. Hospitalization for any reason other than the ACL reconstruction in the last 3 months
5. Plans for additional surgical procedures in the next 12 months
6. Live greater than 60 miles from the research lab
7. Have limitations that would prevent them from attending the biofeedback training sessions
8. Motor neuron diseases, Parkinson's disease, multiple sclerosis
9. Severely impaired hearing or speech (patients must be able to respond to phone calls)
10. No access to a telephone
11. Participating in another ACL intervention
12. Inability to understand or speak English (since this will be required for the patient-based intervention)
13. Other self-reported medical problem that would prohibit participation in the study
14. Other health condition or personal issue judged by a study team member or primary care physician to make the patient inappropriate for study participation
15. Knee extension moment limb symmetry index (LSI) greater than or equal to 90% at the time of the initial study assessment

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin M Queen, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Tech - Kevin P. Granata Biomechanics Lab, Blacksburg, Virginia, United States

REFERENCES:
- [Derived] Peebles AT, Miller TK, Savla J, Ollendick T, Messier SP, Queen RM. Reduction of risk factors for ACL Re-injuries using an innovative biofeedback approach: A phase I randomized clinical trial. Phys Ther Sport. 2022 Sep;57:78-88. doi: 10.1016/j.ptsp.2022.07.007. Epub 2022 Jul 16. PMID 35940085

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Biofeedback Intervention | Control
Started | 18 | 22
Completed | 14 | 22
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biofeedback Intervention | Control | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.2 (1.6) | 16.4 (2.2) | 16.3 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 17 | 19 | 36
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 21 | 35
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 22 | 40
Peak Knee Extension Moment Symmetry [Mean (Standard Deviation); unit: % Symmetry] | 47.9 (28.4) | 41.4 (16.3) | 44.3 (22.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Knee Extension Moment Symmetry
Description: The peak knee extension moment asymmetry will be assessed during the first landing of a stop-jump task
Time Frame: Baseline (week 0) and Post-intervention (week 6)
Population: Analysis completed with participants with >80% adherence
Measure: Mean (Standard Deviation); unit: % Symmetry
Arm/Group | Biofeedback Intervention | Control
Number analyzed (Participants) | 11 | 19
% Symmetry
  Baseline | 50.1 (33.8) | 44.2 (26)
  Post-intervention | 44.6 (24.2) | 40.6 (16.7)

2. Primary Outcome: Change in Peak Knee Extension Moment Symmetry
Description: The peak knee extension moment asymmetry will be assessed during the first landing of a stop-jump task
Time Frame: Post-intervention (week 6) and Retention (week 12)
Population: Analysis completed with participants with >80% adherence
Measure: Mean (Standard Deviation); unit: % Symmetry
Arm/Group | Biofeedback Intervention | Control
Number analyzed (Participants) | 14 | 22
% Symmetry
  Post-intervention | 44.6 (24.2) | 40.6 (16.7)
  Retention | 38.7 (22.5) | 33.3 (13.5)

3. Secondary Outcome: Change in Frontal Plane Knee Range of Motion
Description: The frontal plane knee range of motion will be assessed during the first landing of a stop-jump task
Time Frame: Baseline (week 0) and Post-intervention (week 6)
Population: Analysis completed with participants with >80% adherence
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Biofeedback Intervention | Control
Number analyzed (Participants) | 11 | 19
Degree
  Baseline | 6.4 (2.7) | 10.1 (4.4)
  Post-Intervention | 7.5 (4.5) | 9.1 (4.3)

4. Secondary Outcome: Change in Frontal Plane Knee Range of Motion
Description: The frontal plane knee range of motion will be assessed during the first landing of a stop-jump task
Time Frame: Post-intervention (week 6) and Retention (week 12)
Population: Analysis completed with participants with >80% adherence
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Biofeedback Intervention | Control
Number analyzed (Participants) | 11 | 19
Degree
  Post-intervention | 7.5 (4.5) | 9.1 (4.3)
  Retention | 7.9 (4.2) | 10.1 (4.6)

5. Secondary Outcome: Change in Peak Vertical Ground Reaction Force Symmetry
Description: The peak vertical ground reaction force symmetry will be assessed during the first landing of a stop-jump task
Time Frame: Baseline (week 0) and Post-intervention (week 6)
Population: Analysis completed with participants with >80% adherence
Measure: Mean (Standard Deviation); unit: % Symmetry
Arm/Group | Biofeedback Intervention | Control
Number analyzed (Participants) | 11 | 19
% Symmetry
  Baseline | 34.1 (23) | 28 (9.4)
  Post-intervention | 24.6 (14) | 25.7 (12.9)

6. Secondary Outcome: Change in Peak Vertical Ground Reaction Force Symmetry
Description: The peak vertical ground reaction force symmetry will be assessed during the first landing of a stop-jump task
Time Frame: Post-intervention (week 6) and Retention (week 12)
Population: Analysis completed with participants with >80% adherence
Measure: Mean (Standard Deviation); unit: % Symmetry
Arm/Group | Biofeedback Intervention | Control
Number analyzed (Participants) | 11 | 19
% Symmetry
  Post-intervention | 24.6 (14) | 25.7 (12.9)
  Retention | 32.5 (14.5) | 22.7 (9.2)

ADVERSE EVENTS:
Time Frame: Data was collected over the 12 weeks during which the participants were active on the study.
Arm/Group | Biofeedback Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 0/18 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT03273673/Prot_SAP_000.pdf